CLINICAL TRIAL: NCT02707549
Title: Comparison of Balanced Crystalloid Solution and 0,9% Sodium Chloride in Children Undergoing Brain Tumor Resection: a Randomized Controlled Trial
Brief Title: Fluid Therapy During Brain Tumor Resection in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Mariana Fontes Lima Neville, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 44552315.1.0000.5505
Record Dates: First submitted 2016-03-06; First posted 2016-03-14 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Brain Neoplasms
Keywords: crystalloid solutions; acid-base imbalance; water-electrolyte Imbalance
MeSH Terms: conditions — Brain Neoplasms; Acid-Base Imbalance; Water-Electrolyte Imbalance | interventions — gluconic acid; Sodium Acetate; Potassium Chloride; Magnesium Chloride; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline Group (Active Comparator): the patients included in this group will receive normal saline solution (0.9% sodium chloride) during surgery and in the first 24 hours after ICU admission.
  Interventions: Drug: 0.9% sodium chloride
- Balanced Crystalloid Solution Group (Experimental): the patients included in this group will receive balanced crystalloid solution during surgery and in the first 24 hours after ICU admission.
  Interventions: Drug: balanced crystalloid solution (components: sodium chloride, sodium gluconate, sodium acetate, potassium chloride and magnesium chloride)

INTERVENTIONS:
Drug: balanced crystalloid solution (components: sodium chloride, sodium gluconate, sodium acetate, potassium chloride and magnesium chloride)
  Arms: Balanced Crystalloid Solution Group
Drug: 0.9% sodium chloride
  Arms: Normal Saline Group

SUMMARY:
Fluid management of children during neurosurgery is not well established. Hypotonic solutions, commonly still used in pediatric patients, may enhance cerebral edema and worse operative conditions. This study compares two different isotonic solutions administered perioperatively regarding acid base and fluid electrolyte disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing elective craniotomy for brain tumor resection
* Informed consent form signed and dated by legal guardian and investigator
* Informed assent form signed by the patient if appropriate

Exclusion Criteria:

* Uncontrolled Intracranial hypertension
* Severe heart, kidney, or pulmonary disease
* non-corrected electrolyte imbalance
* allergy to the solution administered

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
serum chloride difference (mmol/L) | from the admission of the patient in the operating room until the end of the surgery.
  Serum chloride will be collected in two different moments: right before the beginning of the surgery and right after de end of the procedure. We will calculate the difference between the two values.

SECONDARY OUTCOMES:
serum chloride difference (mmol/L) | from the end of the surgery until exactly 24 hours after the admission in intensive care unit (ICU)
  Serum chloride will be collected right after the end of the surgery as well as 24 hours after the admission in ICU. We will calculate the difference between the two values.
brain relaxation score | immediately after dura-mater opening
serum sodium difference (mmol/L) | from the admission of the patient in the operating room until the end of the surgery.
  Serum sodium will be collected in two different moments: right before the beginning of the surgery and right after de end of the procedure. We will calculate the difference between the two values.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil